CLINICAL TRIAL: NCT06393816
Title: A Multicenter Phase II Study Evaluating the Efficacy and Safety of the Combination of Durvalumab With Etoposide and Platinum as First Line Treatment in Patients With Large-cell Neuroendocrine Carcinomas (LCNECs) of the Lung
Brief Title: FIRST-NEC (GFPC 01-2022) - Combination of Durvalumab With Etoposide and Platinum
Acronym: FIRST-NEC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET23-132
Record Dates: First submitted 2024-04-17; First posted 2024-05-01 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Large Cell Neuroendocrine Carcinoma of the Lung
Keywords: Advanced; Large Cell Neuroendocrine Carcinoma; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — durvalumab; Etoposide; Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, open-label, phase II study with an external control arm (ESME AMLC database).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental : Durvalumab with etoposide and Carboplatin/Cisplatin (Experimental): Combination of durvalumab with etoposide and platinum (either cisplatin or carboplatin) for the first-line treatment of patients with advanced LCNEC
  Interventions: Drug: Durvalumab with etoposide and Carboplatin/Cisplatin

INTERVENTIONS:
Drug: Durvalumab with etoposide and Carboplatin/Cisplatin — Combination of durvalumab with etoposide and Carboplatin/Cisplatin as First Line Treatment in Patients With Large-cell Neuroendocrine Carcinomas of the Lung.
  All patients (either with confirmed diagnosis or not) will be treated and followed-up:
  * During the induction: every 3 weeks for 12 weeks (4 cycles)
  * During the maintenance: every 4 weeks for 24 months
  Other Names: MEDI4736

SUMMARY:
The primary objective is to determine the efficacy (Progression-Free Rate at 12 months) of durvalumab combined with etoposide and platinum (either cisplatin or carboplatin) for the first-line treatment of patients with advanced LCNEC confirmed by centralized expert-pathologist review

DETAILED DESCRIPTION:
Large-cell neuroendocrine carcinomas (LCNECs) of the lung are lung tumors (2%) included with small-cell lung cancers (SCLCs) in the subgroup of pulmonary neuroendocrine tumors of high-grade malignancy. Histopathological diagnosis of LCNEC is difficult, with a confirmation rate of only 70-80% after centralized expert-pathologist review. The prognosis of advanced LCNECs is poor, with overall survival (OS) of 8-10 months.

The platinum-based regimen is the current recommended first-line treatment for advanced LCNECs in analogy with that given for SCLCs. The previous pivotal GFPC 03-02 trial demonstrated the efficacy of first-line platinum-etoposide in advanced LCNECs with a median Progression-Free Survival (PFS), OS and 1-year PFS of 5 months, 7.7 months and 15% respectively.

The GFPC 03-2017 trial has recently reported that 75% of the tumor samples of LCNEC express programmed cell death protein-ligand-1 (PD-L1) in immune infiltrating tumor cells (ICs), and PD-L1 expression on ICs has been previously correlated with clinical efficacy of Immune Checkpoint Inhibitors (ICI) in Non-small Cell Lung Cancer.

Numerous retrospective studies have also suggested ICI efficacy against LCNECs with significantly prolonged OS observed in ICI-treated LCNEC patients.

Recently, the prospective NIPINEC study results demonstrated second-line nivolumab-ipilimumab efficacy against LCNECs. Moreover, at ESMO 2022, the NICE-NEC prospective phase II study on LCNECs of digestive origin found an impressive efficacy of first-line triplet platinum-etoposide-ICI with a median OS of 13,9 months, and 44 % of long survivor patients (OS>18 months).

Finally, the CASPIAN trial demonstrated the superiority of the combination of durvalumab with platinum-etoposide compared to chemotherapy alone in patients with SCLCs, with an acceptable toxicity profile.

Therefore, within the network of GFPC centers, the investigators propose a prospective, multicenter, open-label, phase II study with an external control arm (ESME database), that aims at evaluating the efficacy and safety of the combination of durvalumab with platinum-etoposide chemotherapy as first-line treatment in patients with an advanced LCNECs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of study entry;
2. Locally documented histological diagnosis of Large-Cell NeuroEndocrine Carcinoma of the lung (2021 WHO classification of Lung Tumors );
3. Patient must have sufficient material to achieve central histological confirmation and exploratory analyses (1 representative FFPE block or at least 10 unstained slides);
4. Setting of the disease: locally advanced (Stage III) not eligible for loco-regional therapy or metastatic (Stage IV) in first line treatment (8th TNM classification).

   Nota Bene: patients with recurrence of local or locally advanced LCNEC are eligible to the trial provided that recurrence occurs beyond 3 months after the last chemotherapy administration.

   For relapsing patients, tumor material collected at diagnosis can be used for the FIRST-NEC trial if relapse occurs within two years of initial management and if initial histologic tumor material is available.
5. Measurable disease as per the RECIST 1.1;
6. Performance Status (PS) of the Eastern Cooperative Oncology Group (ECOG): 0 or 1 ;
7. Body weight > 30Kg;
8. Must have a life expectancy of at least 12 weeks;
9. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥8.0 g/dL (with or without transfusion)
   * Absolute neutrophil count (ANC) ≥1.5 × 109 /L
   * Platelet count ≥100 × 109/L
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN)), or ≤3.0xULN in case of liver metastases.

   Note: this will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
   * For patients undergoing a treatment by cisplatin: measured creatinine clearance (CrCl) ≥60 mL/min or Calculated creatinine CrCl ≥60 mL/min by the CKD-EPI equation or by 24-hour urine collection for determination of creatinine clearance (CrCl).

   Nota Bene: if creatinine clearance is <60 ml/min, patients must be treated with carboplatin rather than cisplatin.
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
11. Patient (male or female) using a highly effective contraception as defined in during the treatment period and at least up to 6 months after the last administration of chemotherapy or 90 days after the last administration of durvalumab, whichever is longer. Prior to dispensing study drugs, the investigator must confirm and document the patient's (and his/her partner) use of highly effective contraceptive methods, dates of negative pregnancy tests, and confirm the patient's understanding of the teratogenic potential of study drugs;
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
13. Affiliation to a social security system;
14. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

1. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study (wash-out period of 28 days);
2. Patient previously treated for a LCNEC in a metastatic setting;
3. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab;
4. Any concurrent chemotherapy, Investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable;
5. Major surgical procedure (as defined by the Investigator) within 21 days prior to the first dose of study drugs; Note: Local surgery or radiotherapy of isolated lesions for palliative intent is acceptable.
6. History of allogenic organ transplantation;
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc).

   The following are exceptions to this criterion:
   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, unstable cardiac arrhythmia, interstitial lung disease, peripheral neuropathy > grade II, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent;
9. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease, or Gleason ≤6 prostate cancer.
10. Central Nervous System metastases, unless asymptomatic (including patients treated with anticonvulsants) or previously treated (surgery or radiation therapy combined with corticosteroids ≤10 mg per day) and stable at the time of randomization for at least 15 days;
11. Carcinomatous meningitis;
12. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms;
13. History of active primary immunodeficiency;
14. Active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA;
15. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection;
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed "10 mg/day" of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.

    Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab.
18. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients;
19. Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
the efficacy (Progression-Free Rate at 12 months) of durvalumab combined with etoposide and platinum (either cisplatin or carboplatin) for the 1st-line treatment of patients with advanced LCNEC confirmed by centralized expert-pathologist review. | 12 months
  The Progression-Free Rate at 12 months (12M-PFR) will be defined as the percentage of patients with a LCNEC confirmed by centralized expert-pathologist review and presenting a complete response (CR), a partial response (PR) or a stable disease (SD) 12 months after the date of treatment start, as per the independent central radiological review committee

SECONDARY OUTCOMES:
12-week Objective Response Rate (ORR) | 12 weeks
  proportion of patients with a LCNEC confirmed by centralized expert-pathologist review with a complete response (CR) or partial response (PR), 12 weeks after the date of treatment start
12-week Disease Control Rate | 12 weeks
  proportion of patients with a LCNEC confirmed by centralized expert-pathologist review with a complete response (CR), partial response (PR) or with stable disease (SD), 12 weeks after the date of treatment start
Progression-Free Survival (PFS) | From date of the first study treatment administration until the date of first documented radiological progression or date of death from any cause, assessed up to 63 months
  time from the date of first study treatment administration to the date of first documented disease progression (reviewed centrally) or the date of death from any cause. Patients without event at the time of analysis will be censored at the date of their last tumor assessment.
Overall Survival | from the date of first study treatment administration to the date of death from any cause, assessed up to 63 months
  time from the date of first study treatment administration to the date of death from any cause. Patients still alive at the time of the analysis will be censored at the time they are known to be alive
Safety profile : description of treatment-emergent Adverse Events | 27 months and 90 days
  All adverse events (AE), all serious adverse events, all immune mediated AE and all Adverse Events of Special Interest will be described using the NCI-CTC version 5.0

OTHER OUTCOMES:
Treatment effectiveness of the experimental combination compared to an external control arm | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 63 months
  PFS and OS will be compared between experimental arm (durvalumab with platinum-etoposide) and an external control arm from the ESME-AMLC real-world database. This comparison will be performed through combined statistical approach using the emulation of a target trial associated with appropriate statistical adjustment techniques to control for confounding biases and thereby reach causal inference capability. The emulation process will consist of outlining key elements of this target trial protocol and then applying them to the ESME data.
Histopathological diagnosis concordance rate | Through central histopathological completion, an average of 6 weeks
  The proportion of patients with a histopathological diagnosis confirmed by central review will be described. The proportion of patients with a histopathological diagnosis confirmed by central review will be described.
12-week Objective Response Rate as a predictive and prognostic factors | 12 weeks
  The 12W-ORR will be studied as predictive (12M-PFR and ORR) and prognostic factors (OS) of efficacy
Overall Survival in the whole study population | From the date of first study treatment administration to the date of death from any cause, assessed up to 63 months
  Overall study as usually published in other studies (in which the diagnosis is not confirmed).
PD-L1 expression as a predictive and prognostic biomarker | From the date of first study treatment administration to the date of death from any cause, assessed up to 63 months
  PD-L1 expression on tumor cells (TCs) and immune cells (ICs), will be studied as predictive (12M-PFR and ORR) and prognostic factors (OS) of efficacy.
Retinoblastoma-1-gene (Rb1) mutation as a predictive and prognostic biomarker | From the date of first study treatment administration to the date of death from any cause, assessed up to 63 months
  Retinoblastoma-1-gene (Rb1) mutation will be studied as predictive (12M-PFR and ORR) and prognostic factors (OS) of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Luc ODIER, MD, Principal Investigator — Hôpital Nord-Ouest, Villefranche sur Saône
Locations (31):
- France (30):
  - Centre Hospitalier Intercommunal Aix-Pertuis, Aix-en-Provence
  - Chu Amiens Picardie Site Sud, Amiens
  - Chu Angers, Angers
  - CENTRE HOSPITALIER d'AVIGNON, Avignon
  - CHU BREST Cavale Blanche, Brest
  - Centre Francois Baclesse, Caen
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Chu Annecy Genevois, Épagny
  - Chu Grenoble Alpes, Grenoble
  - Centre Oscar Lambret, Lille
  - Chu Dupuytren, Limoges
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Centre Leon Berard, Lyon
  - APHM, hôpital nord, Marseille
  - Grand Hopital de L'Est Francilien - Site de Meaux, Meaux
  - GHRMSA, hôpital Emile Muller, Mulhouse
  - CHU NICE, Nice
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - Centre Francois Magendie, Pessac
  - Hospices Civils de Lyon - Lyon Sud Hospital, Pierre-Bénite
  - Centre Hospitalier de Cornouaille, Quimper
  - CHU Rennes, Rennes
  - Institut de Cancerologie Strasbourg Europe, Strasbourg
  - Hopitaux Universitaires de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Hopital Foch, Suresnes
  - Hia Saint Anne, Toulon
  - Chu Toulouse, Toulouse
  - Hopital Nord Ouest de Villefranche Sur Saone, Villefranche-sur-Saône
- Chu Reunion, Réunion, Reunion